CLINICAL TRIAL: NCT05954273
Title: Incidence of Maxillary Sinus Membrane Perforation During Osseodensification Crestal Sinus Grafting
Brief Title: Maxillary Sinus Membrane Perforation Incidence During Osseodensification
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Versah (Industry)
Responsible Party: Sponsor
Other Study IDs: ODSINUSPERF
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Sinus Floor Augmentation; Sinus Infection
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Sinus membrane perforation: Sinus membrane perforation incidences to measure the perforation rate.
  Interventions: Procedure: Osseodensification crestal sinsus graft
- Alveolar bone height below the maxillary sinus floor: Pre-sinus augmentation alveolar bone ridge height.
  Interventions: Procedure: Osseodensification crestal sinsus graft
- Maxillary sinus augementation level: Vertical graft height in the maxillary sinus.
  Interventions: Procedure: Osseodensification crestal sinsus graft
- Implants length and width: Placed implants length and width
  Interventions: Procedure: Osseodensification crestal sinsus graft

INTERVENTIONS:
Procedure: Osseodensification crestal sinsus graft — Osseodensification Mediated Maxillary Sinus Crestal Grafting
  Other Names: Maxillary sinus grafting via crestal approach; Maxillary sinus membrance perforation incidence

SUMMARY:
Measure the incidence of the maxillary sinus membrane perforation during the Osseodensification crestal sinus grafting procedure.

DETAILED DESCRIPTION:
Retrospective clinical study to :

1. Investigate maxillary sinus membrane perforation incidence via osseodensification crestal sinus grafting utilizing the Densah bur.
2. Assess the osseodensification technique efficacy for maxillary crestal sinus grafting with implant site preparation.
3. Study and analyze the maxillary sinus perforation rate during or post-Osseodensification-mediated sinus grafting as a function.
4. To share the knowledge from this retrospective analysis through scientific publications.

ELIGIBILITY:
Inclusion Criteria:

1- Medically healthy patients treated with crestal sinus augmentation via osseodensification using the Densah Burs and implant placement.

Exclusion Criteria:

1. History of radiotherapy,
2. Bisphosphonate medication.
3. Active periodontal disease.
4. Uncontrolled diabetes.
5. Heavy smoking (> 20 cigarettes/day).
6. Local acute apical abscess.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medically healthy patients older than 21 years old who are treated with crestal sinus augmentation via osseodensification using the Densah Burs and implant placement.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-28 (Estimated)

PRIMARY OUTCOMES:
Maxillary sinus membrane perforation rate during osseodensification crestal sinus grafting procedure. | During augmentation surgery
  Measure the incidence of sinus membrane perforation during osseodensification

SECONDARY OUTCOMES:
Maxillary sinus augmentation level | During augmentation surgery
  The height and width of augmentation level

CONTACTS AND LOCATIONS:
Locations (1):
- Versah, LLC, Jackson, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coelho PG, Jimbo R, Tovar N, Bonfante EA. Osseointegration: hierarchical designing encompassing the macrometer, micrometer, and nanometer length scales. Dent Mater. 2015 Jan;31(1):37-52. doi: 10.1016/j.dental.2014.10.007. Epub 2014 Nov 25. PMID 25467952
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329
- [Background] Huwais S, Mazor Z, Ioannou AL, Gluckman H, Neiva R. A Multicenter Retrospective Clinical Study with Up-to-5-Year Follow-up Utilizing a Method that Enhances Bone Density and Allows for Transcrestal Sinus Augmentation Through Compaction Grafting. Int J Oral Maxillofac Implants. 2018 Nov/Dec;33(6):1305-1311. doi: 10.11607/jomi.6770. PMID 30427961
- [Background] Baron Tarun Kumar; Venkatraman Narayan. (2017), Minimally invasive crestal approach sinus floor elevation using Densah burs, and Hydraulic lift utilizing putty graft in cartridge delivery. Clin Oral Impl Res, 28: 203-203.
- [Background] Gaspar, J. , Esteves, T. , Gaspar, R. , Rua, J. and João Mendes, J. (2018), Osseodensification for implant site preparation in the maxilla - a prospective study of 97 implants. Clin Oral Impl Res, 29: 163-163.
- [Background] Alhayati JZ, Al-Anee AM. Evaluation of crestal sinus floor elevations using versah burs with simultaneous implant placement, at residual bone height >/= 2.0 _ < 6.0 mm. A prospective clinical study. Oral Maxillofac Surg. 2023 Jun;27(2):325-332. doi: 10.1007/s10006-022-01071-0. Epub 2022 May 14. PMID 35567659
- [Background] Arafat, Shereen W.; Mohamed A Elbaz. Clinical and radiographic evaluation of Osseodensification versus osteotome for Sinus floor elevation in partially atrophic maxilla: A prospective long term study. Egyptian Dental Journal, 65, issue 1- January (Oral Surgery), 2019, 189-195. Doi: 1021608/edj.2015.71261
- [Background] Neiva R, Tanello B, Duarte W, Silva F. Osseodensification Crestal Sinus Floor Elevation with or without Synthetic and Resorbable Calcium Phosphosilicate Putty. Clin Oral Implants Res. 2018;29 (Suppl.1)
- [Background] Natali C, Ingle P, Dowell J. Orthopaedic bone drills-can they be improved? Temperature changes near the drilling face. J Bone Joint Surg Br. 1996 May;78(3):357-62. PMID 8636166